CLINICAL TRIAL: NCT00241813
Title: Stress Reduction: Impact on Blood Pressure in African American Youth
Brief Title: Effects of Behavioral Stress Reduction Programs on Blood Pressure in African American Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 330; R01HL078216 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Health Education Control Program (CTL) (Active Comparator): Health Education Control Program (CTL)
  Interventions: Behavioral: Health Education Control Program (CTL)
- Mindfulness Meditation (Experimental): Mindfulness Meditation (MM) Program
  Interventions: Behavioral: Mindfulness Meditation (MM) Program
- Lifeskills (Experimental): Lifeskills Program (LP)
  Interventions: Behavioral: Lifeskills Program (LP)
- MM plus LP (Experimental): Mindfulness Meditation (MM) Program plus Lifeskills Program (LP)
  Interventions: Behavioral: Mindfulness Meditation (MM) Program; Behavioral: Lifeskills Program (LP)

INTERVENTIONS:
Behavioral: Mindfulness Meditation (MM) Program — Participants will take part in a mindfulness meditation (MM) program.
  Arms: MM plus LP; Mindfulness Meditation
Behavioral: Health Education Control Program (CTL) — Participants will take part in a health education control program (CTL)
  Arms: Health Education Control Program (CTL)
Behavioral: Lifeskills Program (LP) — Participants will take part in a lifeskills program (LP).
  Arms: Lifeskills; MM plus LP

SUMMARY:
This study will examine the effects of two behavioral stress reduction programs, mindfulness meditation (MM) and the lifeskills program (LP), and a health education control program (CTL) on blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

African Americans (AA) experience a high prevalence and early onset of essential hypertension (EH), which has been partly attributed to exposure to chronic environmental stress. AA youth exhibit higher resting blood pressure (BP) than whites. Since BP ranking tracks from late childhood onward, AA adolescents with high normal BP are at increased risk for development of EH. The need for developing effective primary prevention programs for EH is highlighted by the fact that EH is now a pediatric problem due to recent increased prevalence among youth. There have been no previous controlled studies evaluating stress reduction approaches on BP control in AA youth, particularly within the framework of an underlying psychological and physiological-based model of stress-induced EH.

This study is in response to a 'Request for Applications' entitled "Research on Mind-Body Interactions and Health," which was issued by the Office of the Director, National Institutes of Health (NIH).

DESIGN NARRATIVE:

This study will examine the effects of two behavioral stress reduction programs, MM and LP, and CTL on cardiovascular function at rest, during laboratory stress, and in the natural environment. Participants will include 320 ninth graders (50% male) with high normal systolic BP (SBP) (SBP ranging from greater than or equal to the 50th percentile to less than or equal to the 95th percentile on three occasions). Following BP screenings and baseline evaluation, participants will be assigned to a CTL, MM, LP, or MM plus LP group. Participants will be re-evaluated after a 12-week intervention and again at a 12-week follow-up. The specific aims of this study are to determine whether MM and/or LP results in the following: 1) decreases in the primary outcome variables of resting SBP and 24-hour ambulatory SBP; 2) decreases in sympathetic nervous system (SNS) tone (decreased overnight urine norepinephrine [NE] excretion) and decreases in sodium intake (decreased overnight sodium excretion); 3) decreases in SBP reactivity to behavioral stressors; 4) decreases in SNS arousal (decreased urinary NE excretion) and greater increases in renal function (increased urinary sodium excretion) to the behavioral stressors; 5) decreases in self-reported hostility and anger; 6) improvement in vascular function (increases in percent of endothelium-dependent arterial vasodilation to reactive hyperemia); and 7) improvement in ventricular structure and function (decreases in left ventricular mass index and resting heart rate). It is anticipated that the combination of MM and LP will result in greater positive impacts than either treatment alone. The study will be conducted by teachers during school health classes. If these programs are shown to be successful, they may be incorporated into the regular school curriculum.

ELIGIBILITY:
Inclusion Criteria:

* In ninth grade
* SBP ranging from greater than or equal to 50th percentile to less than or equal to 95th percentile on three occasions

Exclusion Criteria:

* Clinical Hypertension

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Resting SBP and 24-hour ambulatory SBP | Measured after 12-week intervention and at 12-week follow-up

SECONDARY OUTCOMES:
Overnight urine NE excretion | Measured after 12-week intervention and at 12-week follow-up
Overnight sodium excretion | Measured after 12-week intervention and at 12-week follow-up
SBP reactivity to behavioral stressors | Measured after 12-week intervention and at 12-week follow-up
Self-reported hostility and anger | Measured after 12-week intervention and at 12-week follow-up
Percent of endothelium-dependent arterial vasodilation to reactive hyperemia | Measured after 12-week intervention and at 12-week follow-up
Left ventricular mass index and resting heart rate | Measured after 12-week intervention and at 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Treiber, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States